CLINICAL TRIAL: NCT04446312
Title: A Safety and Efficacy Comparison of BLI4900 Bowel Preparation Versus an FDA-approved Comparator in Adult Subjects Prior to Colonoscopy
Brief Title: Study 302: BLI4900 Versus an FDA-approved Comparator in Adult Subjects Prior to Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI4900-302
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLI4900 (Experimental): Experimental bowel preparation solution for oral ingestion
  Interventions: Drug: Bowel Prep
- FDA Approved Control (Active Comparator): FDA approved bowel preparation solution for oral ingestion
  Interventions: Drug: Bowel Prep

INTERVENTIONS:
Drug: Bowel Prep — Orally ingested liquid bowel preparation

SUMMARY:
The purpose of this study is to compare the safety and efficacy of BLI4900 bowel preparation to an FDA-approved control as 2-day, split-dose bowel preparations prior to colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
* 18 to 85 years of age (inclusive)
* If female, and of child-bearing potential, is using an acceptable form of birth control.
* Negative serum pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastroparesis, gastric retention, bowel perforation, toxic colitis or megacolon.
* Subjects with inflammatory bowel disease who have a history of any bowel resection (small intestine or colon), suspected active inflammation, or symptoms suggestive of obstruction or known bowel stricture.
* Subjects who had previous significant gastrointestinal surgeries.
* Subjects who have regularly used laxatives or colon motility altering drugs in the last month (i.e. more than 2-3 times per week) and/or laxative use within 72 hours prior to administration of the preparation
* Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
* Subjects taking diuretics, anti-hypertensive medications, including angiotensin converting enzyme (ACE) inhibitors and Angiotensin II receptor blockers (ARBs), or chronic NSAIDs, that have not been stable for 30 days.
* Subjects with uncontrolled hypertension.
* Subjects taking antibiotics within 7 days of colonoscopy.
* Subjects with severe renal, hepatic or cardiac insufficiency.
* Subjects with an abnormal and clinically significant physical examination or ECG finding at Visit 1.
* Subjects undergoing insulin therapy for any indication.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects undergoing colonoscopy for foreign body removal and/or decompression.
* Subjects taking tricyclic antidepressants.
* Subjects using drugs of abuse, including abused prescription medications.
* Subjects who are withdrawing from alcohol or benzodiazepines.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories / Sebela Pharmaceuticals
Locations (34):
- United States (34):
  - 302 Research Site 2, Tucson, Arizona
  - 302 Research Site 10, Little Rock, Arkansas
  - 302 Research Site 11, North Little Rock, Arkansas
  - 302 Research Site 9, Chula Vista, California
  - 302 Research Site 31, Los Angeles, California
  - 302 Research Site 22, Bristol, Connecticut
  - 302 Research Site 17, Fleming Island, Florida
  - 302 Research Site 3, Inverness, Florida
  - 302 Research Site 14, Jacksonville, Florida
  - 302 Research Site 28, Miami, Florida
  - 302 Research Site 29, Miami, Florida
  - 302 Research Site 30, Miami, Florida
  - 302 Research Site 38, Palm Harbor, Florida
  - 302 Research Site 5, Oak Lawn, Illinois
  - 302 Research Site 34, Baton Rouge, Louisiana
  - 302 Research Site 26, Mandeville, Louisiana
  - 302 Research Site 36, Monroe, Louisiana
  - 302 Research Site 16, Hagerstown, Maryland
  - 302 Research Site 39, Brooklyn, New York
  - 302 Research Site 37, Great Neck, New York
  - 302 Research Site 8, Asheville, North Carolina
  - 302 Research Site 25, High Point, North Carolina
  - 302 Research Site 1, Raleigh, North Carolina
  - 302 Research Site 13, Wilmington, North Carolina
  - 302 Research Site 18, Cincinnati, Ohio
  - 302 Research Site 23, Jackson, Tennessee
  - 302 Research Site 33, Kingsport, Tennessee
  - 302 Research Site 32, Cedar Park, Texas
  - 302 Research Site 21, Houston, Texas
  - 302 Research Site 35, Southlake, Texas
  - 302 Research Site 27, Webster, Texas
  - 302 Research Site 6, Charlottesville, Virginia
  - 302 Research Site 4, Fairfax, Virginia
  - 302 Research Site 7, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhandari R, Goldstein M, Mishkin DS, McGowan J, Cleveland MV, Di Palma JA. Comparison of a Novel, Flavor-optimized, Polyethylene Glycol and Sulfate Bowel Preparation With Oral Sulfate Solution in Adults Undergoing Colonoscopy. J Clin Gastroenterol. 2023 Oct 1;57(9):920-927. doi: 10.1097/MCG.0000000000001894. PMID 37490604

RESULTS

PARTICIPANT FLOW:
Groups:
- BLI4900: Experimental bowel preparation solution for oral ingestion
  Bowel Prep (powder for oral solution): Orally ingested liquid bowel preparation (1 liter per dose)
- FDA Approved Control: FDA approved bowel preparation solution for oral ingestion
  Bowel Prep (liquid for reconstitution): Orally ingested liquid bowel preparation (16 oz per dose)
Period: Overall Study
Arm/Group | BLI4900 | FDA Approved Control
Started | 250 | 250
Completed | 212 | 206
Not Completed | 38 | 44

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population represents the Intent-to-Treat Population which includes all patients that were dispensed a study preparation kit.
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI4900 | FDA Approved Control | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.8) | 56.1 (11.7) | 56.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 152 | 294
  Male | 108 | 98 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 48 | 103
  Not Hispanic or Latino | 195 | 202 | 397
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 11 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 29 | 55
  White | 209 | 213 | 422
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 250 | 250 | 500

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Successful Bowel Preparation
Description: Successful bowel preparation is defined as a preparation rated as Excellent or Good by the blinded endoscopist on a 4 point scale (Excellent, Good, Fair, Poor).
Time Frame: 2 days
Population: Modified intent-to-treat population - this population includes all subjects that took any portion of study preparation and who did not withdraw for a reason other than safety, efficacy or tolerance.
Measure: Count of Participants; unit: Participants
Arm/Group | BLI4900 | FDA Approved Control
Number analyzed (Participants) | 226 | 224
Participants | 212 | 211
Statistical Analysis 1: Comparison: BLI4900 vs FDA Approved Control; Test type: Non-Inferiority — The pre-defined non-inferiority margin was 10%; p < 0.001, Mantel Haenszel; Risk Difference (RD) = 0.15, 95% CI 2-sided [-3.97 to 4.27]

ADVERSE EVENTS:
Time Frame: 30 days
Description: The Analysis Population for adverse event reporting, including serious adverse events and all cause mortality, is the Safety Population which includes all patients that took any portion of the study preparation. This population differs from the Baseline Population because some patients that were dispensed a study preparation did not take it.
Arm/Group | BLI4900 | FDA Approved Control
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/226
Serious Adverse Events (participants affected / at risk) | 0/227 | 2/226
Other Adverse Events (participants affected / at risk) | 23/227 | 26/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI4900 (N=227) | FDA Approved Control (N=226)
concussion (Nervous system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI4900 (N=227) | FDA Approved Control (N=226)
Nausea (Gastrointestinal disorders) | 15 | 14
Vomiting (Gastrointestinal disorders) | 8 | 16
Headache (Nervous system disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT04446312/Prot_SAP_000.pdf